CLINICAL TRIAL: NCT04070690
Title: The Influences of Dialysate Bicarbonate Concentrations on Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Camillians Saint Mary's Hospital Luodong (Other)
Responsible Party: Principal Investigator, Chih-Chung Shiao, MD, Director, Dept. of Medical Research and Education, Saint Mary's Hospital Luodong, Camillians Saint Mary's Hospital Luodong
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SMHRF_107004
Record Dates: First submitted 2019-08-05; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: metabolic acidosis; sodium bicarbonate; hemodialysis; dialysate
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Control group (Other): In this group, the participants will receive "intervention" for 2 months first, followed by a wash-out period of 1 month and "control" for 2 months.
  In the "intervention period," the investigators will provide the participants with lower dialysate HCO3 concentrations. (dialysate HCO3 to 28 mmol/L for half of the HD session and 30 to the second half of their HD session.) Besides, the investigators will give the participants with pre-HD HCO3<22 mEq/L oral Na-bicarbonate 650 mg 1#-2# three times a day as supplements.
  In the "control period," the investigators will provide the participants with dialysate HCO3 concentration of 38-40 mEq/L (as we usually provide to patients).
  Interventions: Procedure: Concentration of dialysate bicarbonate
- Control-Intervention group (Other): In this group, the participants will receive "control" for 2 months first, followed by a wash-out period of 1 month and "intervention" for 2 months.
  In the "control period," the investigators will provide the participants with dialysate HCO3 concentration of 38-40 mEq/L (as we usually provide to patients).
  In the "intervention period," the investigators will provide the participants with lower dialysate HCO3 concentrations. (dialysate HCO3 to 28 mmol/L for half of the HD session and 30 to the second half of their HD session.) Besides, the investigators will give the participants with pre-HD HCO3<22 mEq/L oral Na-bicarbonate 650 mg 1#-2# three times a day as supplements.
  Interventions: Procedure: Concentration of dialysate bicarbonate

INTERVENTIONS:
Procedure: Concentration of dialysate bicarbonate — Adjust the dialysate bicarbonate concentration

SUMMARY:
Background:

Patients with decreased kidney function are in the positive acid balance due to insufficient renal acid excretion. To correct the varying degrees of metabolic acidosis in these HD patients, a high concentration of HCO3 in the dialysate is routinely used.

During every 3-to-4 hours of HD treatment, a massive surge of HCO3 would enter the circulation and typically overcorrects predialysis acidosis to alkalosis and alkalemia.

The sharp acid-base shift can cause some adverse consequences.

The investigators believe that the rapid correction (or overcorrection) from the pre-dialysis metabolic acidosis to post-dialysis metabolic alkalosis during the 3-to-4 hours HD treatment would relate to adverse effects on HD patients.

Thus the investigators conduct this study to prove the hypothesis that "prevention of post-dialysis alkalosis by using lower dialysate HCO3 concentration might cause less adverse outcomes in ESRD patients on HD."

Study design:

Prospective cross-over case-control study.

Study population:

A total of 60 patients who receive regular hemodialysis (three times per week) for more than 6 months in the regional teaching hospital.

ELIGIBILITY:
Inclusion Criteria:

* adult uremic patients who received hemodialysis thrice weekly

Exclusion Criteria:

* Hospitalized patients
* Patients newly initiated on HD (<6 months)
* Patients with HD access problems
* Patients recently discharged from the hospital (within one month).
* Patients on chemotherapy for cancer.
* Patients with a kidney transplant.
* Patients on steroids or other immunosuppressive therapy.
* Patients with recent surgery (within one month)
* Patients with an active bacterial infection.
* Patients with decompensated cirrhosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Blood pressure during the hemodialysis | four months
  Blood pressure will be measured every 1 hour during the hemodialysis
Respiratory rate during the hemodialysis | four months
  Respiratory rate will be measured every 1 hour during the hemodialysis
O2 saturation during the hemodialysis | four months
  O2 saturation will be measured every 1 hour during the hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chung Shiao, MD, Principal Investigator — Saint Mary's Hospital Luodong
Locations (1):
- Saint Mary's Hospital Luodong, Yilan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The influences of dialysate bicarbonate concentrations on hemodialysis patients